CLINICAL TRIAL: NCT03090893
Title: A Pilot Study, Prospective, Non-Randomized, Non-Blinded, Single-Center Study Evaluating the Response of Continuous Recombinant Antithrombin (ATryn) Infusion in Postcardiotomy ECMO Patients
Brief Title: Response of Continuous Recombinant Antithrombin Infusion in Postcardiotomy ECMO Patients
Status: Withdrawn | Phase: Early Phase 1 | Type: Interventional
Why Stopped: PI passed away
Sponsor: Mayo Clinic (Other)
Collaborators: rEVO Biologics (Industry)
Responsible Party: Principal Investigator, William C. Oliver, PI, Mayo Clinic
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: 15-001713
Record Dates: First submitted 2017-03-21; First posted 2017-03-27 (Actual); Last update posted 2018-09-10 (Actual); Status verified 2018-09

CONDITIONS: Antithrombin Deficiency Type 2
MeSH Terms: conditions — Antithrombin deficiency type 2

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (1):
- Infusion group (Experimental): Subjects will receive ATryn continuous infusion for maintaining serum antithrombin III levels between 80 - 100
  Interventions: Drug: ATryn continuous infusion

INTERVENTIONS:
Drug: ATryn continuous infusion — replenish serum thrombin levels

SUMMARY:
The objective of this study will be to prospectively evaluate the response of a continuous infusion of recombinant human antithrombin concentrate (rhAT) (ATRYN®) to achieve and maintain the AT activity within a specified range in adult patients that require extracorporeal membrane oxygenation (ECMO) following cardiopulmonary bypass (CPB) and cardiac surgery.

ELIGIBILITY:
Inclusion Criteria:

* Completed cardiac surgery with Cardiopulmonary Bypass and subsequently placed on venoarterial (VA) Extracorporeal Membrane Oxygenation (ECMO) support at any point during the ongoing hospitalization
* Serum Antithrombin < 60%.

Exclusion Criteria:

* Heart transplantation during ongoing hospitalization
* Excessive bleeding (300 ml/hr of chest tube drainage for 2 consecutive hours)
* Weight < 40 kg
* Allergy to goat products
* Anticoagulation with a direct thrombin inhibitor
* Religious exception to blood products
* Hypothermia (< 34°C)

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2018-06-01 (Estimated); Primary Completion 2019-06 (Estimated); Study Completion 2019-06 (Estimated)

PRIMARY OUTCOMES:
Percentage of time within the serum AT level target range of 80-100% | 72 hour infusion period
  Target value of Antithrombin is recorded as %

CONTACTS AND LOCATIONS:
Overall Officials: William C. Oliver, Jr., MD, Principal Investigator — Mayo Clinic

IPD SHARING:
Plan to Share IPD: No
will not share individual patient data